CLINICAL TRIAL: NCT04990310
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-CORT113176 in Healthy Male Subjects
Brief Title: Single Dose Absorption, Distribution, Metabolism, and Excretion Study of [14C]-CORT113176 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CORT113176-651; 2021-002544-78 (EudraCT Number)
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): On Day 1, participants will receive a single oral dose of [14C]-CORT113176 450 mg (3 X 150 mg lipid formulation capsules) in the fed state.
  Interventions: Drug: [14C]-CORT113176

INTERVENTIONS:
Drug: [14C]-CORT113176 — [14C]-CORT113176 450 mg lipid formulation capsule for oral administration containing not more than 3.37 megaBequerel 14C.

SUMMARY:
This study will evaluate the mass balance recovery and metabolite profile, and will identify metabolite structures following a single oral dose of [14C]-CORT113176 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 30.0 kg/m^2, inclusive
* Willing and able to participate in the whole study
* Have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day)
* Provide written informed consent
* Adhere to the contraception requirements.

Exclusion Criteria:

* Have received any investigational medicine in a clinical research study within 90 days
* Are, or are immediate family members of, a study site or sponsor employee
* Evidence of current severe acute respiratory syndrome (SARS-CoV-2) infection
* History of any drug or alcohol abuse, or regularly consume >21 units alcohol per week
* Current smoker or user of e-cigarettes and nicotine replacement products within the last 6 months
* Have pregnant or lactating partners
* Radiation exposure, exceeding 5 milliSieverts (mSv) in the last 12 months or 10 mSv in the last 5 years
* Clinically significant abnormal results of clinical chemistry, hematology or urinalysis as judged by the investigator
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* Active renal and/or hepatic disease
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal (GI) disease, neurological or psychiatric disorder
* Any form of cancer within the last 5 years (exceptions apply)
* History and/or symptoms of adrenal insufficiency
* Condition that could be aggravated by glucocorticoid antagonism or activation
* Donation of blood or plasma or loss of greater than 400 mL of blood within the previous 3 months
* Are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) within 14 days. COVID-19 vaccines are accepted concomitant medications. Exceptions may apply on a case by case basis.
* Currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months or 3 months for inhaled products
* Additional criteria apply.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Mass Balance Recovery in Excreta After a Single Dose of [14C]-CORT113176 | Until the mass balance criteria for all participants have been met (estimated up to 28 days)

SECONDARY OUTCOMES:
Mass Balance Recovery in Urine After a Single Oral Dose of [14C]-CORT113176 | Until the mass balance criteria for all participants have been met (estimated up to 28 days)
Mass Balance Recovery in Feces After a Single Oral Dose of [14C]-CORT113176 | Until the mass balance criteria for all participants have been met (estimated up to 28 days)
Number of CORT113176 Metabolites Accounting for ≥10% of Total Circulating Radioactivity or ≥10% of Dose Excreted in Urine and Feces | Until the mass balance criteria for all participants have been met (estimated up to 28 days)
Plasma Pharmacokinetics (PK) of Total Radioactivity after Oral Dosing: Peak Plasma Concentration (Cmax) | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Time from Dosing to Cmax (Tmax) | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Area Under the Plasma Concentration-time Curve from Zero Time to Time of the Last Measurable Concentration (AUC0-last) | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Apparent Elimination Half-life (t1/2) | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT113176 after Oral Dosing: Cmax | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT113176 after Oral Dosing: Tmax | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT113176 after Oral Dosing: AUC0-last | Before dosing and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT113176 after Oral Dosing: t1/2 | Before dosing and at pre-specified time points up to Day 8 after dosing
Distribution of Total Radioactivity into Red Blood Cells after Oral Dosing | Before dosing and at pre-specified time points up to Day 8 after dosing
Number of Participants with One or More Adverse Events | Until the mass balance criteria for all participants have been met (estimated up to 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Hunt, Ph.D., Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No